CLINICAL TRIAL: NCT02230813
Title: Prevalence and Predictors of Initial Oral Antibiotic Treatment Failure in Adult Emergency Department Patients With Cellulitis: a Pilot Study
Brief Title: Predictors of Oral Antibiotic Treatment Failure in Emergency Department Patients With Cellulitis
Status: Completed | Type: Observational
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Other Study IDs: 14/53
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Cellulitis
Keywords: Cohort Study,; Cellulitis,; Skin and Soft Tissue Infection,; Emergency Department,; Clinical Prediction Rule
MeSH Terms: conditions — Cellulitis; Soft Tissue Infections; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Oral antibiotic therapy: Consecutive adult patients attending the study Emergency Departments with cellulitis will be considered eligible for recruitment to the study. Only those patients deemed suitable for oral antibiotic therapy and planned for discharge will be recruited to the study. Oral antibiotic therapy prescribed will be dependent on local institutional prescribing guidelines. For the purposes of the sites enrolling participants, the antibiotic of choice is oral flucloxacillin 500 milligrams four times daily for seven days. We will be assessing the treatment failure rate for this cohort of patients; namely, the number of patients requiring the primary outcome (change from oral to intravenous antibiotic therapy). We will also assess this group of patient for the secondary outcomes listed above.

SUMMARY:
The term cellulitis is a medical term describing a bacterial infection of the skin and tissues beneath the skin. Although it is usually easily treated with antibiotics given either orally or through a vein (intravenously), knowing which route of antibiotic treatment to prescribe to a person attending an Emergency Department with cellulitis is not clear.

A Clinical Prediction rule (CPR) is a decision-making tool that comes from original research as opposed to the opinion of experts. We intend to create a preliminary CPR to decide which patients require oral and which patients require intravenous antibiotics for cellulitis from their first visit to an emergency department. The aim of this is to provide safer care by reducing the risk of a patient returning to the hospital with a worsening infection. It will also promote more cost-effective care by reducing hospital re-attendance rates and wasted antibiotics.

Patients attending the department with cellulitis who are suitable for oral antibiotic treatment will be enrolled into this study. A separate doctor will re-examine at least 10% of study participants in order to reduce bias. A set of physical signs and symptoms will be recorded from each patient in order to determine which ones are associated with them "failing" prescribed oral treatment. A study investigator will then phone the patient after 14 days to see whether they are better or whether they required intravenous antibiotics to get better.

ELIGIBILITY:
Inclusion Criteria:

* Age >16 years
* Suitable for treatment with flucloxacillin 500mg -1gram qds monotherapy or a suitable alternative for penicillin allergic patients as listed in the local prescribing guidelines.
* Appearance of typical, plaque-like area of erythema over any body part excluding the perineum within the preceding 5 days with any 2 of the following signs:
* 1.Increased warmth over affected area
* 2.Swelling of affected area
* 3.Pain over affected area
* 4.Regional lymphadenopathy

Exclusion Criteria:

* Requirement for IV antibiotics as decided by the treating clinician.
* Age less than 16 years.
* No telephone or access to a telephone.
* Abscess alone without co-existing signs of cellulitis
* Mammalian bite wounds.
* Infected diabetic foot ulcer
* Necrotising soft tissue infections.
* Perineal cellulitis.
* Suspected septic arthritis or osteomyelitis.
* Decubitus ulcers.
* Bilateral cellulitis (as this entity rarely exists).
* Acute lipodermatosclerosis.
* Acute dermatitis.
* Venous stasis dermatitis.
* Deep vein thrombosis.
* Pregnancy.
* Cognitive impairment.
* Any patient who through language barrier or diminished capacity is unable to understand the scope of the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients aged >16 years attending the ED with cellulitis as the primary diagnosis will be consecutively recruited. Only patients who are deemed suitable for an oral antibiotic will be enrolled. Patients who require IV therapy will not be enrolled. Cellulitis may arise de novo, or from a recognised cause such as a wound or ulcer. In order to generate an externally valid clinical prediction rule, we will include all patients attending the ED with cellulitis, including those who may have already been commenced on oral antibiotics (for example, by their general practitioner).
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09-27 (Actual); Study Completion 2016-09-27 (Actual)

PRIMARY OUTCOMES:
Treatment failure | 2 weeks post commencement of oral treatment
  The primary outcome is the proportion of patients initially commenced on oral antibiotics who subsequently require IV antibiotics to achieve treatment response. This will be assessed by means of telephone follow-up performed at 14 days post enrolment into the study. Treatment failure is defined as attendance at a treating Emergency Department for intravenous antibiotic therapy if already commenced on oral therapy.

SECONDARY OUTCOMES:
Treatment failure - change in type or dose | 2 weeks
  Treatment failure measured by change in prescribed oral antibiotic to another oral antibiotic.
  Treatment failure measured by change in prescribed dose of oral antibiotic to a higher dose of the same antibiotic
Inter-observer reliability for candidate predictor variables | At enrolment
  Assessment of inter-observer reliability for the candidate predictor variables listed. This will be performed in at least 10% of patients enrolled into the study by a second recruiting clinician.
Loss to follow up | 2 weeks
  Assessment of the loss to follow-up rate and usefulness of the data collection proforma in the pilot study will also prove valuable for planning for the live study.

CONTACTS AND LOCATIONS:
Overall Officials: Abel Wakai, MD FRCS FCEM, Principal Investigator — Royal College of Surgeons, Ireland
Locations (3):
- Ireland (3):
  - Connolly Hospital Banchardstown, Dublin
  - Emergency Department Beaumont Hospital, Dublin
  - Mater Misericoridiae University Hospital, Dublin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Quirke M, Mitchell N, Varley J, Kelly S, Boland F, Moughty A, McKeever J, Fahey T, Wakai A. Prevalence and predictors of oral to intravenous antibiotic switch among adult emergency department patients with acute bacterial skin and skin structure infections: a pilot, prospective cohort study. BMJ Open. 2020 Aug 30;10(8):e034057. doi: 10.1136/bmjopen-2019-034057. PMID 32868346
- [Derived] Quirke M, Boland F, Fahey T, O'Sullivan R, Hill A, Stiell I, Wakai A. Prevalence and predictors of initial oral antibiotic treatment failure in adult emergency department patients with cellulitis: a pilot study. BMJ Open. 2015 Jun 25;5(6):e008150. doi: 10.1136/bmjopen-2015-008150. PMID 26112223